CLINICAL TRIAL: NCT07019129
Title: Effects of Dietary Nitrate in Women With Secondary Amenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Coggan, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 26781
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Secondary Amenorrhea
Keywords: dietary nitrate; secondary amenorrhea; muscle function
MeSH Terms: interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Nitrate-free beetroot juice
  Interventions: Dietary Supplement: Placebo Beetroot Juice Without Nitrate
- Nitrate (Experimental): Nitrate-rich beetroot juice
  Interventions: Dietary Supplement: Beetroot Juice - Active

INTERVENTIONS:
Dietary Supplement: Beetroot Juice - Active — Nitrate-rich beetroot juice
  Arms: Nitrate
Dietary Supplement: Placebo Beetroot Juice Without Nitrate — Nitrate-poor beetroot juice
  Arms: Placebo

SUMMARY:
Excessive exercise, disordered attitudes toward eating, physical and psychological stress, and/or hormonal imbalances may result in cessation of menstruation (secondary amenorrhea). The accompanying lack of estrogen may impair muscle power and oxygen recovery after exercise by reducing nitric oxide levels. The purpose of this study is to determine whether ingestion of beetroot juice containing nitrate, an alternative source of nitric oxide, can help reverse these changes.

DETAILED DESCRIPTION:
Due to excessive exercise, disordered attitudes toward eating, physical and psychological stress, and/or hormonal imbalances, young women may be predisposed to developing secondary amenorrhea. Secondary amenorrhea is defined as the absence of menses for at least 3 months in regularly menstruating women or at least 6 months in irregularly menstruating women [1]. This disorder of the hypothalamic-pituitary axis (HPO) is associated with a short-term lack of endogenous estradiol (E2), which may have negative health consequences [2-7]. For example, E2 plays an important role in regulating skeletal muscle mass and contractile function, including both strength and power [4]. In part, this is because E2 increases phosphorylation of the regulatory light chain of myosin, thereby enhancing muscle contractility [6, 8]. Lack of E2 also alters lipid and carbohydrate metabolism [9, 10], which may be due to the important role E2 plays in regulating mitochondrial function, more specifically respiration and efficiency. This impairment in metabolism and mitochondrial respiration could increase CVD risk and alter plasma levels of lipids, cortisol, and insulin [2, 9, 10]. Indeed, Ronkainen et al. [11] found that postmenopausal women not on hormone replacement therapy (HRT) have reduced skeletal muscle strength and power compared to those on HRT, whereas Kleis-Olsen et al. [12] reported similar findings with respect to fat mass and mitochondrial respiratory capacity. Younger women with secondary amenorrhea may also suffer from similar impairments due to E2 deficiency.

It has also been shown that short term lack of E2 compromises nitric oxide synthase (NOS) activity, which plays a critical role in cardiovascular health, exercise capacity, and vasomodulation and mitochondrial function within skeletal muscle [7, 13, 14]. Conversely, dietary nitrate supplementation can increase nitric oxide bioavailailbity, via an enterosalivary pathway in which nitrate is reduced to nitrite that in turn is further reduced to nitric oxide [15]. It has been demonstrated that dietary nitrate improves muscle contractility [16], exercise capacity and performance [15, 17], vascular function [18], and mitochondrial efficiency during exercise [5, 19, 20]. Indeed, we have found nitrate supplementation to be particularly effective in increasing muscular speed and power in postmenopausal women [21]. Increasing NO bioavailability via ingestion of nitrate therefore may have beneficial effects on both muscle function and mitochondrial function in women with secondary amenorrhea. To date, however, this hypothesis has not been tested.

Although the aforementioned research has highlighted the beneficial effects of dietary nitrate supplementation on muscle contractile function and mitochondrial respiration in various populations, no studies have examined the effects of this supplementation on these parameters in women with secondary amenorrhea. The proposed study will therefore provide a better understanding of the effects of dietary nitrate supplementation on muscle function and mitochondrial respiration in women with secondary amenorrhea, potentially improving health, recovery, and performance outcomes within this vulnerable population.

1. Rebar, R., Evaluation of Amenorrhea, Anovulation, and Abnormal Bleeding, in Endotext, K.R. Feingold, et al., Editors. 2000: South Dartmouth (MA).
2. Gupte, A.A., H.J. Pownall, and D.J. Hamilton, Estrogen: an emerging regulator of insulin action and mitochondrial function. J Diabetes Res, 2015. 2015: p. 916585.
3. Ihalainen, J.K., et al., Beyond Menstrual Dysfunction: Does Altered Endocrine Function Caused by Problematic Low Energy Availability Impair Health and Sports Performance in Female Athletes? Sports Med, 2024. 54(9): p. 2267-2289.
4. Chidi-Ogbolu, N. and K. Baar, Effect of Estrogen on Musculoskeletal Performance and Injury Risk. Front Physiol, 2018. 9: p. 1834.
5. Larsen, F.J., et al., Dietary inorganic nitrate improves mitochondrial efficiency in humans. Cell Metab, 2011. 13(2): p. 149-59.
6. Lai, S., et al., Estradiol modulates myosin regulatory light chain phosphorylation and contractility in skeletal muscle of female mice. Am J Physiol Endocrinol Metab, 2016. 310(9): p. E724-33.
7. O'Donnell, E. and M.J. De Souza, The cardiovascular effects of chronic hypoestrogenism in amenorrhoeic athletes: a critical review. Sports Med, 2004. 34(9): p. 601-27.
8. Greenberg, M.J., et al., The molecular effects of skeletal muscle myosin regulatory light chain phosphorylation. Am J Physiol Regul Integr Comp Physiol, 2009. 297(2): p. R265-74.
9. An, J., et al., Sex- and endurance training-mediated cardiovascular protection through lipids during exercise. Trends Endocrinol Metab, 2024.
10. Senoz, S., et al., Estrogen deprivation, rather than age, is responsible for the poor lipid profile and carbohydrate metabolism in women. Maturitas, 1996. 25(2): p. 107-14.
11. Ronkainen, P.H., et al., Postmenopausal hormone replacement therapy modifies skeletal muscle composition and function: a study with monozygotic twin pairs. J Appl Physiol (1985), 2009. 107(1): p. 25-33.
12. Kleis-Olsen, A.S., et al., Metabolic flexibility in postmenopausal women: Hormone replacement therapy is associated with higher mitochondrial content, respiratory capacity, and lower total fat mass. Acta Physiol (Oxf), 2024. 240(6): p. e14117.
13. Fadel, P.J., W. Zhao, and G.D. Thomas, Impaired vasomodulation is associated with reduced neuronal nitric oxide synthase in skeletal muscle of ovariectomized rats. J Physiol, 2003. 549(Pt 1): p. 243-53.
14. Tengan, C.H., G.S. Rodrigues, and R.O. Godinho, Nitric oxide in skeletal muscle: role on mitochondrial biogenesis and function. Int J Mol Sci, 2012. 13(12): p. 17160-84.
15. Amdahl, M.B., A.W. DeMartino, and M.T. Gladwin, Inorganic nitrite bioactivation and role in physiological signaling and therapeutics. Biol Chem, 2019. 401(1): p. 201-211.
16. Coggan, A.R. and L.R. Peterson, Dietary Nitrate Enhances the Contractile Properties of Human Skeletal Muscle. Exerc Sport Sci Rev, 2018. 46(4): p. 254-261.
17. Flueck, J.L., et al., Is beetroot juice more effective than sodium nitrate? The effects of equimolar nitrate dosages of nitrate-rich beetroot juice and sodium nitrate on oxygen consumption during exercise. Appl Physiol Nutr Metab, 2016. 41(4): p. 421-9.
18. Craig, J.C., et al., Effect of dietary nitrate supplementation on conduit artery blood flow, muscle oxygenation, and metabolic rate during handgrip exercise. J Appl Physiol (1985), 2018. 125(2): p. 254-262.
19. Bailey, S.J., et al., Dietary nitrate supplementation enhances muscle contractile efficiency during knee-extensor exercise in humans. J Appl Physiol (1985), 2010. 109(1): p. 135-48.
20. Pappas, G., M.L. Wilkinson, and A.J. Gow, Nitric oxide regulation of cellular metabolism: Adaptive tuning of cellular energy. Nitric Oxide, 2023. 131: p. 8-17.
21. Coggan, A.R., et al., Dietary nitrate-induced increases in human muscle power: high versus low responders. Physiol Rep, 2018. 6(2).
22. Jungersten, L., et al., Plasma nitrate as an index of nitric oxide formation in man: analyses of kinetics and confounding factors. Clin Physiol, 1996. 16(4): p. 369-79.
23. Govoni, M., et al., The increase in plasma nitrite after a dietary nitrate load is markedly attenuated by an antibacterial mouthwash. Nitric Oxide, 2008. 19(4): p. 333-7.
24. Joint FAO/WHO Expert Committee on Food Additives. Meeting (61st: 2003, R., Italy) & International Programme on Chemical Safety., Safety evaluation of certain food additives and contaminants/prepared by the sixty-first meeting of the Joint FAO/WHO Expert Committee on Food Additives (JEFCA). 2004.
25. Goodman, J., S. Thomas, and J.F. Burr, Physical activity series: cardiovascular risks of physical activity in apparently healthy individuals: risk evaluation for exercise clearance and prescription. Can Fam Physician, 2013. 59(1): p. 46-9, e6-e10.
26. Sumner, M.D., et al., Near Infrared Spectroscopy Measurements of Mitochondrial Capacity Using Partial Recovery Curves. Front Physiol, 2020. 11: p. 111.
27. Gallardo EJ, Gray DA, Hoffman RL, Yates BA, Moorthi RN, Coggan AR. Dose-response effect of dietary nitrate on muscle contractility and blood pressure in older subjects: a pilot study. J Gerontol A Biol Sci Med Sci 2021; 76:591-598.
28. Zoughaib WS, Hoffman RL, Yates BA, Moorthi RN, Lim K, Coggan AR. Short-term beetroot juice supplementation improves muscle contractility but does not reduce blood pressure or oxidative stress in 65-79 y old men and women. Nitric Oxide 20

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-44 years old
* Missed >3 consecutive periods in the last 12 months if previously regularly menstruating (average cycle 21-35 d) OR
* Missed >6 consecutive periods in the last 12 month if previously irregularly menstruating (spontaneous menstruation, average cycle <21 or > 35 d)

Exclusion Criteria:

* Unable to provide informed consent
* Currently diagnosed with primary amenorrhea (no history of menstruation by age 15) or oligomenorrhea (menstrual cycle >35 d or <8 cycles per year)
* Currently diagnosed with a chronic illness, including thyroid disease, hyperprolactinemia, Cushing syndrome, and/or poly-cystic ovarian syndrome (PCOS)
* History or current clinical diagnosis of an eating disorder
* Currently dieting
* Weight instablility for the past 3 months
* Previously undergone a revascularization procedure involving a vascular graft or stenting of the femoral or popliteal arteries
* Currently at the time of screening, or in the past year, using hormonal contraceptives
* Pregnancy
* Epilepsy
* Current antibiotic use
* Current nicotine user
* Stage II hypertension (resting blood pressure >140/>90)
* Currently taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy
* An answer of yes to any of the seven questions on the first page of the Physical Activity Readiness Questionnaire (PAR-Q) indicating that the participant is not physically ready for exercise without a medical exam. These exclusions include the following:
* If participant's doctor has ever said that he/she has a heart condition and that he/she should only do physical activity recommended by a doctor
* Pain in chest when doing physical activity
* In past month, chest pain when not doing physical activity
* If participant has ever lost balance because of dizziness or has ever lost consciousness
* Muscle, bone, or joint problem that could be made worse by physical activity
* Currently on prescribed drugs for blood pressure or heart condition.
* If the participant knows of any other reason he/she should not do physical activity.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximal knee extensor power | Approximately 2-3 hours after beetroot ingestion
  Maximal power of the knee extensor (thigh) muscles as determined using isokinetic dynamometry
Muscle reoxygenation kinetics | Approximately 2-3 hours after beetroot juice ingestion
  Recovery rate constant (k) of muscle oxygenation following exercise as determined using NIRS (near-infrared spectroscopy) combined with brief intermittent arterial occlusion

SECONDARY OUTCOMES:
Maximal knee extensor velocity | Approximately 2-3 hours after beetroot juice ingestion
  Maximal velocity of the knee extensor (thigh) muscles as determined using isokinetic dynamometry
Deoxygenation rate | Approximately 2-3 hours after beetroot juice ingestion
  Rate of deoxygenation of the knee extensor (thigh) muscles during 5 minutes of continuous arterial occlusion as determined using NIRS (near-infrared spectroscopy)
Reoxygenation rate | Approximately 2-3 hours after beetroot juice ingestion
  Rate of reoxygenation of the knee extensor (thigh) muscles following 5 minutes of continuous arterial occlusion as determined using NIRS (near-infrared spectroscopy)

OTHER OUTCOMES:
Baseline plasma nitrate/nitrite concentration | Before beetroot juice ingestion
  Concentrations of nitrate and nitrite in blood plasma as determined using HPLC (high performance liquid chromatography)
Plasma nitrate/nitrite concentration at 1 hour | 1 hour after beetroot juice ingestion
  Concentrations of nitrate and nitrite in blood plasma as determined using HPLC (high performance liquid chromatography)
Plasma nitrate/nitrite concentration at 2 hours | 2 hours after beetroot juice ingestion
  Concentrations of nitrate and nitrite in blood plasma as determined using HPLC (high performance liquid chromatography)
Plasma nitrate/nitrite concentration at 3 hours | Approximately 3 hours after beetroot juice ingestion
  Concentrations of nitrate and nitrite in blood plasma as determined using HPLC (high performance liquid chromatography)
Estradiol concentration | Before beetroot juice ingestion
  Concentration of estradiol (E2) in blood plasma as determined using ELISA (enzyme linked immunosorbent assay)
Follicle stimulating hormone concentration | Before beetroot juice ingestion
  Concentration of follicle stimulating hormone (FSH) in blood plasma as determined using ELISA (enzyme linked immunosorbent assay)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Coggan, PhD, Principal Investigator — Indiana University Indianapolis
Locations (1):
- Indiana University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-PHI individual participant data will be shared upon reasonable request.
Time Frame: Data will be made available upon completion of the study and publication of the final results.